CLINICAL TRIAL: NCT04673357
Title: A Phase 3 Study of the Efficacy, Safety, and Pharmacokinetics of Ustekinumab as Open-label Intravenous Induction Treatment Followed by Randomized Double-blind Subcutaneous Ustekinumab Maintenance in Pediatric Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Ustekinumab in Pediatric Participants With Moderately to Severely Active Crohn's Disease
Acronym: UNITI Jr
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108864; CNTO1275CRD3004 (Other: Janssen Research & Development, LLC); 2019-004225-24 (EudraCT Number); 2023-504978-38-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease
Keywords: Pediatric
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Induction period is an open-label period and maintenance period is a double-blind period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open- Label Ustekinumab Intravenous (IV): Induction Period (Experimental): All participants will receive a single IV administration of ustekinumab at induction Week 0 (I-0) based on body surface area (BSA) (milligram per meter square [mg/m^2]) or weight-tiered induction dose (milligram per kilogram [mg/kg]).
  Interventions: Drug: Ustekinumab
- Ustekinumab Subcutaneous (SC) Every 8 Weeks (q8w): Maintenance Period (Experimental): Participants will receive SC administration of ustekinumab q8w based on BSA (mg/m^2) or weight-tiered induction dose (mg/kg) at maintenance weeks (Weeks M)-0, M-8, M-16, M-24, M 32, and M-40 and matching placebo at Weeks M-12 and M-36 to maintain the blind.
  Interventions: Drug: Ustekinumab; Drug: Placebo
- Ustekinumab SC Every 12 Weeks (q12w): Maintenance Period (Experimental): Participants will receive SC administration of ustekinumab q12w based on BSA (mg/m^2) or weight-tiered induction dose (mg/kg) at Weeks M-0, M-12, M-24, M-36 and matching placebo at Weeks M-8, M-16, M-32, and M-40 to maintain the blind.
  Interventions: Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab will be administered intravenously in induction period and subcutaneously in maintenance period.
Drug: Placebo — Matching placebo will be administered as SC injection.
  Arms: Ustekinumab SC Every 12 Weeks (q12w): Maintenance Period; Ustekinumab Subcutaneous (SC) Every 8 Weeks (q8w): Maintenance Period

SUMMARY:
The purpose of this study is to evaluate the efficacy of ustekinumab dosing in inducing clinical remission (Global) and in maintaining clinical remission (US); to evaluate the safety profile and ustekinumab exposure (pharmacokinetics [PK]) in pediatric participants with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease or fistulizing Crohn's disease with active colitis, ileitis, or ileocolitis, confirmed at any time in the past by endoscopy and histology
* Must have moderately to severely active Crohn's disease (as defined by a baseline Pediatric Crohn's Disease Activity Index [PCDAI] score greater than [>] 30); have ileocolonoscopy with evidence of active Crohn's disease defined as presence of ulceration (which is equal to Simple Endoscopic Score for Crohn's disease [SES-CD] score greater than or equals to [>=] 3) during screening into this study. The ileocolonoscopy procedure must occur within approximately 3 weeks prior to the administration of study intervention at Week 0 (Induction Period). A video ileocolonoscopy recorded within 3 months prior to the Week 0 (Induction Period) visit may be used in case of rescreening of a participant who had an ileocolonoscopy but failed the initial screening for another reason, on a case-by-case basis, after consultation with the sponsor. If unable to evaluate ulceration due to stricture or inadequate bowel preparation, at least one of the following criteria may instead be applied: an abnormal C-reactive protein (CRP) (> 0.3 milligram per deciliter [mg/dL] or 3.0 milligram per liter [mg/L] at screening) or; fecal calprotectin of >= 250 milligram per kilogram [mg/kg] or >= 250 microgram per gram [mcg/g] at screening
* If receiving enteral nutrition, must have been on a stable regimen for at least 2 weeks prior to induction week 0 (Week I-0)
* Females of childbearing potential must have a negative highly sensitive urine pregnancy test at screening and at Week I-0 prior to study intervention administration

Exclusion Criteria:

* Has complications of Crohn's disease such as symptomatic strictures or stenosis, short gut syndrome, or any other manifestation that might be anticipated to require surgery, that could preclude the use of the PCDAI to assess response to therapy or would possibly confound the ability to assess the effect of treatment with ustekinumab
* Have a history of latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis, or have had a nontuberculous mycobacterial infection prior to screening
* Presence or history of any malignancy including presence or history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (example, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic areas), and monoclonal gammopathy of undetermined significance, or clinically significant hepatomegaly or splenomegaly
* Have a history of moderate or severe progressive or uncontrolled liver or renal insufficiency; or significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric (including suicidality), or metabolic disturbances
* Received an investigational intervention including any investigational vaccines or used an invasive investigational medical device within 3 months before the planned first dose of study intervention or is currently enrolled in an investigational study; receipt of an investigational vaccine for Coronavirus Disease 2019 (COVID-19) is not an automatic exclusion criterion

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Clinical Remission at Induction Week 8 | Week 8
  Number of participants with clinical remission in induction period will be assessed. Clinical remission is defined as having a Pediatric Crohn's Disease Activity Index (PCDAI) score less than or equal to (<=) 10 points. PCDAI is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdominal tenderness or mass, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease.
Number of Participants with Adverse Events (AEs) | Up to Week 74
  An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | Up to Week 74
  A SAE is any untoward medical occurrence that at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with AEs leading to Discontinuation of Study Intervention | Up to Week 74
  Number of participants with AEs leading to discontinuation of study intervention will be reported.
Number of Participants with AEs of Interest | Up to Week 74
  Number of participants with AEs of interest (any newly identified malignancy, or case of active tuberculosis [TB], or opportunistic infection occurring after the first administration of study intervention[s]) will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to Week 52
  Number of participants with abnormalities in clinical laboratory parameters (such as hematology and chemistry) will be reported.
Number of Participants with Reactions Temporally Associated with Intravenous (IV) Infusion (Induction Period) | Up to Week 8 (Induction period)
  Number of participants with reactions temporally associated with IV infusion in induction period will be reported.
Number of Participants with Subcutaneous (SC) Injection-Site Reactions (Maintenance Period) | Up to Week 44 (Maintenance period)
  Number of participants with SC injection-site reactions in maintenance period will be reported.
Serum Ustekinumab Concentrations | Up to Week 52
  Serum ustekinumab concentrations will be reported.
Number of Participants with Clinical Remission at Maintenance Week 44 | Week 44 (Maintenance Period)
  Number of participants with clinical remission in maintenance period will be assessed. This will be assessed among participants who are in clinical response at induction week-8 (I-8). Clinical remission is defined as having a PCDAI score <= 10 points. PCDAI is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdominal tenderness or mass, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease.

SECONDARY OUTCOMES:
Number of Participants with Clinical Remission as Assessed by short Pediatric Crohn's Disease Activity Index (sPCDAI) | Week 6 (Induction period)
  Number of participants with clinical remission in induction period as assessed by sPCDAI will be reported. Clinical remission is defined as PCDAI score and sPCDAI score <= 10 points.
Number of Participants with Clinical Response | Week 8 (Induction period)
  Number of participants with clinical response in induction period will be reported.
Number of Participants with Clinical Response as Assessed by sPCDAI | Week 6 (Induction period)
  Number of participants with clinical response in induction period as assessed by sPCDAI will be reported. Clinical response is defined as a reduction from baseline in the PCDAI score of greater than or equal to (>=) 12.5 points with a total PCDAI score not more than 30.
Number of Participants with Endoscopic Response as Assessed by Simplified Endoscopic Score-Crohn's Disease (SES-CD) | Week 8 (Maintenance period)
  Number of participants with endoscopic response as assessed by SES-CD in maintenance period will be reported. Endoscopic response is defined as a reduction in SES-CD score of >= 50 percent (%) or SES-CD score <= 2 in participants with a baseline SES-CD score of >= 3. The SES-CD score is based on the evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component is scored from 0 to 3 for each segment, and a total score is derived from the sum of all the component scores (range, 0 to 60).
Number of Participants with Clinical Response | Week 8 (Maintenance period)
  Number of participants with clinical response in maintenance period will be reported.
Number of Participants with Clinical Remission | Week 44 (Maintenance period)
  Number of participants with clinical remission in maintenance period will be reported.
Number of Participants with Endoscopic Response as Assessed by SES-CD | Week 44 (Maintenance period)
  Number of participants with endoscopic response as assessed by SES-CD in maintenance period will be reported. Endoscopic response is defined as a reduction in SES-CD score of >= 50 percent (%) or SES-CD score <= 2 in participants with a baseline SES-CD score of >= 3. The SES-CD score is based on the evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component is scored from 0 to 3 for each segment, and a total score is derived from the sum of all the component scores (range, 0 to 60).
Number of Participants with Clinical Response | Week 44 (Maintenance period)
  Number of participants with clinical response in maintenance period will be reported.
Number of Participants with Corticosteroid-free Clinical Remission | Week 44 (Maintenance period)
  Number of participants with corticosteroid-free clinical remission in maintenance period will be reported. Corticosteroid-free clinical remission is PCDAI score <= 10 points and not receiving corticosteroids for at least 90 days prior to Week 44.
Number of Participants with Clinical Remission at Week 44 (Maintenance Period) who are in Clinical Remission at Week 8 (Induction Period) | Week 44 (Maintenance Period)
  Number of participants with clinical remission at Week 44 (maintenance period) who are in clinical remission at Week 8 (induction period) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (9):
  - Nemours DuPont Hospital for Children, Wilmington, Delaware
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Levine Childrens at Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Cook Childrens Medical Center, Fort Worth, Texas
  - Pediatric Specialists Of Virginia, Fairfax, Virginia
- Belgium (5):
  - Universitair Kinderziekenhuis Koningin Fabiola, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
- Germany (7):
  - Universitätsklinikum Aachen, Aachen
  - Charite-Universitätsmedizin Berlin - Berlin, Berlin
  - Universitatsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Dr. von Haunersches Kinderspital, Munich
  - KUNO Klinik St. Hedwig, Regensburg
  - Universitatsklinikum Ulm, Ulm
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod Abauj Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szabolcs Szatmar Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Szegedi Tudományegyetem, Gyermekgyógyászati Klinika és Gyermekegészségügyi Centrum, Szeged
- Israel (4):
  - Yitzhak Shamir Medical Center, Be’er Ya‘aqov
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
- Japan (9):
  - Juntendo University Hospital, Bunkyō City
  - Gunma University Hospital, Gunma
  - Kindai University Nara Hospital, Ikoma
  - Kurume University Hospital, Kurume
  - Saitama Childrens Medical Center, Saitama Shi
  - Miyagi Children's Hospital, Sendai
  - National Center for Child Health and Development, Setagaya Ku
  - Jichi Medical University Hospital, Shimotsuke
  - Mie University Hospital, Tsu
- Poland (5):
  - Szpital im. M. Kopernika, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Russia (4):
  - Kazan State Medical University, Kazan'
  - Russian National Research Medical University named after N.I.Pirogov, Moscow
  - Privolzhsky Research Medical University of Ministry of Health of Russian Federation, Nizhny Novgorod
  - Yaroslavl Regional Children's Clinical Hospital, Yaroslavl
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Hospital for Children and Young People, Edinburgh
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency